CLINICAL TRIAL: NCT00083590
Title: A Multi-Center, Double-Blind, Placebo-Controlled Therapeutic Trial to Determine Whether Natural Huperzine A Improves Cognitive Function
Brief Title: Huperzine A in Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Alzheimer's Disease Cooperative Study (ADCS) (Other); Neuro-Hitech (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IA0052; ADC-023; IND 63,997
Record Dates: First submitted 2004-05-26; First posted 2004-05-27 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2008-02

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; Cholinesterase inhibitor
MeSH Terms: conditions — Alzheimer Disease | interventions — huperzine A

INTERVENTIONS:
Drug: Huperzine A

SUMMARY:
The present study will evaluate the safety and efficacy of the Chinese herb huperzine A in the treatment of Alzheimer's disease (AD) in a randomized controlled trial of its effect on cognitive function.

DETAILED DESCRIPTION:
Huperzine A is a natural cholinesterase inhibitor derived from the Chinese herb Huperzia serrata. There is evidence that huperzine A may compare favorably in symptomatic efficacy to cholinesterase inhibitors currently in use. In addition, huperzine A has antioxidant and neuroprotective properties that suggest that it may be useful as a disease-modifying treatment for Alzheimer's disease (AD). The drug is currently available as a nutraceutical in this country, and is being used by some U.S. clinicians to treat AD. However, there have been no controlled clinical trials outside China assessing its toxicity and efficacy. The present study will evaluate huperzine A in the treatment of AD in a randomized controlled trial of its effect on cognitive function.

The primary aim of this multicenter, double-blind, placebo-controlled therapeutic Phase II trial is to determine whether treatment with huperzine A 200µg twice a day improves cognitive function in individuals with AD. Secondary aims of this study are to: a) determine whether treatment with huperzine A 400µg twice a day improves cognitive function in individuals with AD; b) determine the effect of huperzine A treatment on global clinical status, activities of daily living, and behavior in AD; c) evaluate the tolerability of huperzine A treatment at dosages of 200µg twice a day and 400µg twice a day in AD; and d) determine the relationship between blood cholinesterase activity and cognitive function in individuals with AD treated with huperzine A. A total of 150 participants will be randomly assigned to three groups of equal size. This will allow a comparison of huperzine A 200µg twice a day, huperzine A 400µg twice a day, and placebo. The primary outcome measures will be the change in score on the ADAScog at the 16 week visit. Secondary outcome measures include the ADCS clinical global impression of change (CGIC) (Schneider et al 1997) and activities of daily living (ADL) (Galasko et al 1997) scales, and the Neuropsychiatric Inventory (Cummings 1997). Volunteers must be able to participate in the study for 24 weeks and make 9 visits to the trial site.

At the end of the double-blind study, participants will be invited to continue huperzine A treatment for 6 months in an open-label extension phase. Participants will receive 200µg of huperzine A twice a day for six consecutive months, and will be assessed at 3-month intervals (months 6, 9, and 12, with month 6 assessments coinciding with the final visit of the double-blind phase).

ELIGIBILITY:
The selection process is designed to allow enrollment of all people with AD who are likely to be testable at the conclusion of the study period, and who do not have concurrent medical conditions or medications that might influence cognitive testing or that would increase the risk of treatment. Women and members of minority groups are encouraged to volunteer.

Inclusion Criteria:

* NINDS/ADRDA criteria for probable AD.
* Mini Mental State Examination between 10 and 24, inclusive.
* Stable medical condition for 3 months prior to screening.
* Supervision available for administration of study medications.
* Study partner to accompany participant to all scheduled visits.
* Fluent in English or Spanish.
* Age 55 years or older.
* Modified Hachinski score equal to or less than 4.
* CT or MRI since onset of memory impairment demonstrating absence of clinically significant focal lesion.
* Able to complete baseline assessments.
* 6 years of education, or work history sufficient to exclude mental retardation.
* Able to ingest oral medication.
* Stable doses of medications for 4 weeks prior to screening.
* Physically acceptable for this study as confirmed by medical history, physical exam, neurological exam and clinical tests.

Exclusion Criteria:

* History of active peptic ulcer disease within 1 year of screening.
* Clinically significant cardiac arrhythmia.
* Resting pulse less than 50.
* Active neoplastic (cancer) disease (skin tumors other than melanoma are not excluded; participants with stable prostate cancer may be included at the discretion of the Project Director).
* Use of another investigational agent within 2 months of screening.
* History of clinically significant stroke.
* Current evidence or history in the past 2 years of epilepsy, focal brain lesion, head injury with loss of consciousness and/or immediate confusion after the injury, or DSM-IV criteria for any major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse.
* Blindness, deafness, language difficulties or any other disability which may prevent the participant from participating or cooperating in the protocol.
* Residence in a skilled nursing facility; but patients in an assisted living facility are acceptable.

Excluded Medications:

* Use of cholinesterase inhibitors (galantamine, rivastigmine, donepezil, and tacrine) within 2 months of screening.
* Regular use of narcotic analgesics (>2 doses per week) within 4 weeks of screening.
* Use of medications with significant central nervous system anticholinergic activity within 2 months of screening (e.g. tricyclic antidepressants, diphenhydramine).
* Use of anti-Parkinsonian medications (including Sinemet, amantadine, bromocriptine, pergolide, selegiline) within 2 months of screening.
* Participation in any other investigational drug study within 2 months of screening (individuals may not participate in any other drug study while participating in this protocol).
* Use of estrogen is allowed if the dose has been stable for 3 months prior to screening.
* Use of vitamin E is allowed if the dose has been stable for 3 months prior to screening.
* Use of memantine is allowed if the dose has been stable for 3 months prior to screening.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2004-04; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul S. Aisen, MD, Principal Investigator — Georgetown University Medical Center, Memory Disorders Program
Locations (29):
- United States (29):
  - University of Alabama, Birmingham, Alabama
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - University of California, Irvine, Irvine, California
  - University of California, San Diego, Alzheimer's Disease Research Center, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - Georgetown University Medical Center, Memory Disorders Program, Washington D.C., District of Columbia
  - Howard University School of Medicine, Washington D.C., District of Columbia
  - MD Clinical, Fort Lauderdale, Florida
  - Roskamp Institute Memory Clinic, Tampa, Florida
  - University of South Florida, Suncoast Alzheimer's and Gerontology Center, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Rush Alzheimer's Disease Center, Rush University Medical Center, Chicago, Illinois
  - ICPS Group, Boston, Massachusetts
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - Alzheimer's Research Corporation, Paterson, New Jersey
  - University of Medicine and Dentistry of New Jersey, Piscataway, New Jersey
  - Albany Medical Center, Albany, New York
  - New York University Medical Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Nathan S. Kline Institute for Psychiatric Research, Orangeburg, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, North Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Vermont College of Medicine, Burlington, Vermont

REFERENCES:
- [Background] Bai DL, Tang XC, He XC. Huperzine A, a potential therapeutic agent for treatment of Alzheimer's disease. Curr Med Chem. 2000 Mar;7(3):355-74. doi: 10.2174/0929867003375281. PMID 10637369
- [Background] Ved HS, Koenig ML, Dave JR, Doctor BP. Huperzine A, a potential therapeutic agent for dementia, reduces neuronal cell death caused by glutamate. Neuroreport. 1997 Mar 3;8(4):963-8. doi: 10.1097/00001756-199703030-00029. PMID 9141073
- [Background] Mazurek A: An open-label trial of huperzine A in the treatment of Alzheimer's disease. Alternative Therapies 5(2): 97-98, March 16, 2000.